CLINICAL TRIAL: NCT03855462
Title: Evaluating Efficacy and Safety of Medium-chain Triglycerides Used as a Temporary Intraocular Tamponading Agent for Retinal Detachment Treated by Endocular Surgery
Brief Title: Evaluating Medium-chain Triglycerides as a Temporary Intraocular Tamponading Agent for Retinal Detachment
Acronym: MCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0360
Record Dates: First submitted 2018-12-05; First posted 2019-02-26 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Ophthalmopathy
Keywords: endotamponade; retinal detachment; vitreoretinal proliferation
MeSH Terms: conditions — Eye Diseases; Retinal Detachment | interventions — Mucociliary Clearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCT oil injection (Experimental): The patient treatment is the classical surgical procedure which is used for retinal detachment with silicon oil medium-chain triglycerides (MCT) as tamponade agent :
  * Vitrectomy, then flattened retina, and finally MCT injection in place of the vitreous.
  * MCT ablation after 4 to 6 weeks (after effective retinopexy)
  Interventions: Device: MCT oil injection

INTERVENTIONS:
Device: MCT oil injection — The patient treatment is the classical surgical procedure which is used for retinal detachment with MCT oil :
  * Vitrectomy, then flattened retina, and finally MCT injection in place of the vitreous.
  * MCT ablation after 4 to 6 weeks (after effective retinopexy)
  * after MCT ablation, total follow-up duration by patient is 6 months.

SUMMARY:
Background : Surgery is needed in order to flatten and position a detached retina onto the choroid, to allow sealing of the tears and to prevent or reverse vision loss. In case of complex retinal detachment vitrectomies followed by ocular endotamponade - non-solid implants used in ophthalmology - is the most common treatment. Despite several options used by surgeons were not entirely satisfactory, no innovation were marketed in the ocular endotamponade field since decades.

Purpose : Regarding comparative physico-chemical properties of medium-chain triglycerides (MCT) with current tamponading agents (silicone oil or gases), it will be proposed to evaluate the MCT as an ocular endotamponade product.

DETAILED DESCRIPTION:
Previously a nonclinical study has provide an assessment of the safety and the local tissue effects of the Medium-Chain Triglyceride (MCT) tamponade agent manufactured by the company Arcadophta : There were no histopathologic findings or irritation events that were directly attributable to the MCT device. In conclusion, under the conditions of the study, the MCT device did not induce any adverse local tissue effects compared to a control tamponading agent silicone oil.

The present clinical study is the first use of MCT tamponade agent which assigns human participants. The MCT tamponade agent studied is manufactured by the company Arcadophta and designed as a Class IIb medical device in Europe.

Tamponment efficacy and human eye safety of the device are supported by a flatten retina observation and a healthy eye fundus exam respectively as long as the tamponade agent is present.

The patient treatment is the classical surgical procedure which is used for retinal detachment with silicone oil.

* Vitrectomy, then flattened retina, and finally MCT injection in place of the vitreous.
* MCT ablation after 4 to 6 weeks (after effective retinopexy) The patient follow-up begins 4 days before treatment , then 3 time-points exams are performed before MCT ablation and 4 time-points exams are performed after MCT ablation for a total patient follow-up duration of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Each patient with retinal detachment which requires a classical surgical procedure with silicone oil.
* Proliferative vitreoretinopathy over C2 regarding Retina Society classification
* Retinal detachment due to trauma to the eye
* Retinal detachment due to equatorial wound dehiscence which requires a classical surgical procedure with silicone oil.
* Retinal detachment due to complex proliferative diabetic retinopathy
* Recurrence of retinal detachment after ophthalmic gaz treatment
* Retinal detachment due to giant tear (>90°C independently of the location into the eye.

Exclusion Criteria:

* monophthalmic patient
* Eye with corneal dystrophy
* Intraocular pressure > 25 mmHg under treatment
* Patient with travel difficulty or living place far away from the clinic
* Patient participating to another clinical study.
* Pregnant women or breastfeeding women
* Patient under tutors or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Efficacy (tamponment efficacy supported by a flatten retina observation) | 6 month
  Flatten retina observation by fundus exam

SECONDARY OUTCOMES:
Efficacy (injection facility of MCT oïl) | Inclusion day : Day 0
  Facility injection of MCT oil as tamponment assessed according to a 4-point scale (from 0=very easy to 3=very difficult)
Efficacy (ablation facility of MCT oïl) | 6 weeks
  Facility ablation of MCT oil assessed according to a 4-point scale (from 0=very easy to 3=very difficult)
Safety (MCT emulsification) | 6 month
  MCT emulsification assessed according to 5-point scale (from grade 0 = absence of emulsification to grade 4= emulsification that not allow to distinguish retinal details, unobservable fundus
presence of micro-bubbles after post MCT ablation assessed according to a 5-point scale | 6 month
  Safety secondary outcomes is evaluate by presence of micro-bubbles post MCT ablation according to 5-point scale (from grade 0 = absence of emulsification to grade 4= emulsification that not allow to distinguish retinal details, unobservable fundus
Presence of hypertonia (intraocular pressure) | 6 month
  The presence of hypertonia will be assessed by measurement of the intraocular pressure. An ocular hypertonia is defined by an intraocular pressure superior to 25 mmHg
Safety (Inflammation) | 6 month
  Presence of inflammation in the anterior chamber (Tyndall) or in the vitreous cavity according to the ophthalmic examination
Cataract presence (lens opacity classification system III) | 6 month
  The presence or worsening of cataract will be assessed according to the lens opacity classification system III
Keratopathy presence to evaluate safety of MCT oil | 6 month
  Presence of keratopathy will be assessed using a 4-point scale (from 0 = absence to 3 = keratopathy with strips)
distance visual acuity measure to evaluate safety of MCT oil | 6 month
  Safety secondary outcomes is evaluated by distance visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Pagot-Mathis, MD, Principal Investigator — CHU of Toulouse, FRANCE
Locations (2):
- France (2):
  - Polyclinique Saint Roch, Montpellier
  - University Hospital Toulouse (Hospital Pierre Paul Riquet), Toulouse

IPD SHARING:
Plan to Share IPD: No